CLINICAL TRIAL: NCT06864715
Title: Behavioral Activation for the PreVention of Post-strokE Depression in LoW-incomE Older Stroke Survivors (LIVE-WEL)
Brief Title: Behavioral Activation for the PreVention of Post-strokE Depression in LoW-incomE Older Stroke Survivors
Acronym: LIVE-WEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Beauchamp, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SN-25-XXXX
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Post-stroke Depression; Subthreshold Depression
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-delivered Behavioral Activation by lay counselors after Stroke (Tele-BA-S) (Experimental)
  Interventions: Behavioral: Tele-delivered Behavioral Activation by lay counselors after Stroke (Tele-BA-S)
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Tele-delivered Behavioral Activation by lay counselors after Stroke (Tele-BA-S) — The Tele-BA-S intervention will comprise 5 weekly video-conferenced BA sessions delivered by trained lay counselors, homework, and 2 monthly follow-up booster calls.
  Arms: Tele-delivered Behavioral Activation by lay counselors after Stroke (Tele-BA-S)
Behavioral: Treatment as Usual — Participants will receive an educational packet and blood pressure (BP) monitor prior to hospital discharge. They will be contacted by a Licensed Clinical Social Worker (LCSW) at 48-72 hours to determine if they have received their medications and appointments. The stroke practitioner will evaluate patients at 7-14 days and 3 months ±14 days, according to current standard of care. They will be seen over video or in-person, according to their preference and capabilities.
  Arms: Treatment as Usual

SUMMARY:
The overall objective of the project is to determine the effectiveness of tele-delivered behavioral activation (BA) by trained lay counselors (Tele-BA-S) to prevent Post-stroke depression (PSD) in low-income, older stroke survivors with subthreshold depression (SD).

DETAILED DESCRIPTION:
Post-stroke depression (PSD) affects an estimated 33% of survivors. Subthreshold depression (SD; clinically relevant depressive symptoms that do not meet diagnostic criteria for a clinical disorder) can affect up to 60% of stroke survivors and, if untreated, likely progresses to PSD. PSD is associated with recurrent stroke, mortality (including suicide), neurological deficits, and diminished functioning and quality of life (QOL). Older survivors are at particularly high risk for PSD owing to age-related life stressors (e.g., chronic disabilities and conditions, polypharmacy, bereavement, and dependence on others). For low-income, older stroke survivors, financial strain is an added risk factor for PSD. Treating SD may prevent PSD. However, first-line pharmacological treatment for PSD prevention can be problematic for older survivors who may fear dependency and can be sensitive to adverse effects and drug-drug interactions. Behavioral activation (BA) is an efficacious depression treatment that increases engagement in value-based, reinforcing activities and decreases avoidance behaviors. BA does not require licensed therapists, is less costly and as effective as cognitive therapy for reducing depression, and can be modified to effectively target behaviors that have been empirically associated with risk for PSD. The overall objective of the proposal is to determine the effectiveness of tele-delivered BA by trained lay counselors (Tele-BA-S) to prevent PSD in low-income, older stroke survivors with SD. A randomized controlled trial will be conducted (Tele-BA-S vs. treatment-as-usual [TAU]; n=280) with follow-up at 2-months, 4-months, 6-months, and 9-months after baseline to test the short- and long-term effectiveness of Tele-BA-S. Participants will be low-income, older (≥ 55 years) first-time ischemic or hemorrhagic survivors (≤ 6 months after stroke) with SD. The intervention will comprise 5 weekly video-conferenced BA sessions delivered by trained lay counselors, homework, and 2 monthly follow-up booster calls. Aim 1 is to test the effectiveness of Tele-BA-S vs. TAU on reducing symptoms of SD and the proportion of survivors that develop PSD (primary clinical outcome). Aim 2 is to test the effectiveness of Tele-BA-S vs TAU on reducing anxiety, emotional distress, and healthcare visits and improving QOL and disability (secondary outcomes). Aim 3 is to investigate self-efficacy, motivation, and activity engagement as mediators of Tele-BA-S effectiveness for reducing symptoms of SD and the proportion of survivors that develop PSD.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment within 6-months of a first-time ischemic or hemorrhagic stroke
* 24-item HDRS score between 5 to 8 indicating the presence of mild symptoms of depression
* Single person income less than or equal to $45,000
* Residing in a community residence
* Ability to speak and read in English or Spanish

Exclusion Criteria:

* Stroke event unrelated to vascular risk factors (e.g., drug use) or transient ischemic attack
* 24-item HDRS score > 8 indicating moderate to severe depression
* Actively participating in psychotherapy
* high suicide risk or severe psychiatric illness (e.g., bipolar disorder and active psychosis)
* Diagnosed dementia
* Diagnosed aphasia, visual, and/or severe cognitive impairments [Montreal Cognitive Assessment (MoCA) score ≤ 17]

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-Stroke Depression as Assessed by Score on the Hamilton Depression Rating Scale (HDRS) 24-item | baseline, 2 months, 4 months, 6 months, 9 months
  Total score on the 24-item HDRS ranges from 0 to 15, with a higher score indicating greater depression, as follows:
  * 0-4: normal
  * 5-8: mild
  * 8-11: moderate
  * 12-15: severe
Subthreshold Depression as Assessed by the Patient Health Questionnaire (PHQ-9) | baseline, 1 month, 2 months, 4 months, 6 months, 9 months
  Total score on the PHQ-9 ranges from 0 to 27, with a higher score indicating greater depression, as follows:
  * 5-9: mild depression
  * 10-14: moderate depression
  * 15-19: moderately severe depression -≥ 20: severe depression

SECONDARY OUTCOMES:
Anxiety as Assessed by the Generalized Anxiety Disorder- 7 Item (GAD-7) | baseline, 2 months, 4 months, 6 months, 9 months
  Total score on the GAD-7 ranges from 0 to 15, with a higher score indicating greater anxiety, as follows:
  * 0-4: Minimal Anxiety
  * 5-9: Mild Anxiety
  * 10-14: Moderate Anxiety -≥ 15: Severe Anxiety
Emotional Distress as Assessed by the General Health Questionnaire-28 (GHQ-28) | baseline, 2 months, 4 months, 6 months, 9 months
  Total score on the GHQ-28 ranges from 0 to 84, with a higher score indicating higher levels of distress.
Quality of Life (QOL) as Assessed by the Stroke Specific Quality of Life Scale (SS-QOL) | baseline, 2 months, 4 months, 6 months, 9 months
  Total score on the SS-QOL ranges from 49-245, with a higher score indicating better functioning.
Number of Self-Reported Emergency Room Visits Over the Course of the Study | From baseline to 9 months
Number of Hospitalizations Over the Course of the Study | From baseline to 9 months
Disability as Assessed by the Modified Rankin Scale (mRS) | baseline, 2 months, 4 months, 6 months, 9 months
  Total score on teh mRS ranges from 0-6, with a higher score indicating greater disability, as follows:
  * 0: No symptoms at all
  * 1: No significant disability despite symptoms; able to carry out all usual duties and activities
  * 2: Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  * 3: Moderate disability; requiring some help, but able to walk without assistance
  * 4: Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  * 5: Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  * 6: Dead

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Beauchamp, PhD, RN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No